CLINICAL TRIAL: NCT00666679
Title: Randomized, Placebo-controlled Clinical Trial to Study the Efficacy and Safety of Inhaled Corticosteroid Plus Montelukast Compared With Inhaled Corticosteroid Therapy Alone in Patients With Chronic Asthma
Brief Title: Study of Inhaled Corticosteroid Plus Montelukast Compared With Inhaled Corticosteroid Therapy Alone in Patients With Chronic Asthma (0476-386)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-386; MK0476-386; 2007_654
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2010-02-03 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): mometasone
  Interventions: Drug: Comparator: mometasone
- 2 (Placebo Comparator): montelukast followed by placebo; or placebo followed by montelukast.
  Interventions: Drug: Comparator: montelukast; Drug: Comparator: placebo (unspecified)

INTERVENTIONS:
Drug: Comparator: mometasone — mometasone (inhalation powder, 220 mcg once-daily, for approximately 6 weeks)
  Arms: 1
Drug: Comparator: montelukast — montelukast (inhalation powder, 1 mg once-daily, for approximately 2 weeks)
  Arms: 2
Drug: Comparator: placebo (unspecified) — Placebo (Placebo once-daily, for approximately 2 weeks)
  Arms: 2

SUMMARY:
This study assesses inhaled corticosteroid plus montelukast compared with inhaled corticosteroid therapy alone for treatment of patients with chronic asthma.

DETAILED DESCRIPTION:
During this study, all patients will receive mometasone (powder, 220 mcg once-daily, for approximately 6 weeks). In a crossover manner, eligible patients will also receive montelukast (powder, 1 mg once-daily, for approximately 2 weeks) followed by placebo; or will receive placebo followed by montelukast. The order of when each of these 2 treatments are added to the mometasone will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Patient has decreased breathing capacity (when not taking asthma medicine) that improves after taking a fast-acting asthma inhaler
* Within one month of the first study visit, patient has been treated with a fast-acting asthma inhaler, and may be treated with a corticosteroid inhaler or an inhaler that combines a corticosteroid plus a bronchodilator

Exclusion Criteria:

* Patient is hypersensitive to inhaled beta-agonists, corticosteroids, leukotriene antagonists, or any of their components
* Has required an oral corticosteroid rescue for worsening asthma during the screening period

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Philip G, Villaran C, Shah SR, Vandormael K, Smugar SS, Reiss TF. The efficacy and tolerability of inhaled montelukast plus inhaled mometasone compared with mometasone alone in patients with chronic asthma. J Asthma. 2011 Jun;48(5):495-502. doi: 10.3109/02770903.2011.573042. Epub 2011 May 5. PMID 21545249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 25 centers worldwide. Patient screening began 05-May-2008 and the first patient was randomized on 29-May-2008.
  The last patient's last visit was completed on 16-Feb-2009.
Pre-assignment Details: 278 participants were screened; 144 were excluded.
  Randomized patients met the following criteria: FEV1 (Forced expiratory volume in one second) 50-80% predicted while withholding short-acting beta agonist (SABA) and reversibility of airway obstruction >12% following SABA documented on at least two of the following visits: Visits 1, 2, and 3.
Groups:
- Montelukast + Mometasone Then Placebo + Mometasone: Patients were randomized to receive montelukast 1 mg (milligram) and open-label mometasone 220 mcg (micrograms) once daily by inhalation in the first intervention; and placebo for montelukast and open-label mometasone 220 mcg once daily by inhalation in the second intervention (after washout). During washout, patients received open-label inhaled mometasone 220 mcg and single-blind placebo for montelukast once daily by inhalation.
- Placebo + Mometasone Then Montelukast + Mometasone: Patients were randomized to receive placebo for montelukast and open-label mometasone 220 mcg once daily by inhalation in the first intervention; and montelukast 1 mg and open-label mometasone 220 mcg once daily by inhalation in the second intervention (after washout). During washout, patients received open-label inhaled mometasone 220 mcg and single-blind placebo for montelukast once daily by inhalation.
Period: First Intervention
Arm/Group | Montelukast + Mometasone Then Placebo + Mometasone | Placebo + Mometasone Then Montelukast + Mometasone
Started | 66 | 68
Completed | 62 | 67
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Randomized did not start treatment | 1 | 1
Period: Washout Period of 1 Week
Arm/Group | Montelukast + Mometasone Then Placebo + Mometasone | Placebo + Mometasone Then Montelukast + Mometasone
Started | 62 | 67
Completed | 62 | 65
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Second Intervention
Arm/Group | Montelukast + Mometasone Then Placebo + Mometasone | Placebo + Mometasone Then Montelukast + Mometasone
Started | 62 | 65
Completed | 61 | 64
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast + Mometasone Then Placebo + Mometasone | Placebo + Mometasone Then Montelukast + Mometasone | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (15.5) | 42.6 (14.8) | 40.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 69
  Male | 29 | 36 | 65
Daytime Asthma Symptom Score (0 [best] to 6 [worst] Point Scale) [Mean (Standard Deviation); unit: Units on a Scale] | 2.04 (0.90) | 2.18 (0.81) | 2.11 (0.85)
FEV1 (Forced Expiratory Volume in One Second) [Mean (Standard Deviation); unit: L (Liter)] | 2.14 (0.67) | 2.18 (0.55) | 2.16 (0.61)
Nighttime Asthma Symptom Score (0 [best] to 3 [worst] Point Scale) [Mean (Standard Deviation); unit: Units on a Scale] | 0.51 (0.53) | 0.46 (0.48) | 0.49 (0.50)
Total Daily Beta-Agonist Use [Mean (Standard Deviation); unit: Puffs] | 3.52 (2.49) | 3.55 (2.19) | 3.53 (2.34)
Total Peripheral Blood Eosinophils [Mean (Standard Deviation); unit: 10^3/microliters] | 0.46 (0.39) | 0.38 (0.31) | 0.42 (0.35)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in FEV1 (Forced Expiratory Volume; Volume of Air That is Exhaled During the First Second of a Forced Exhalation)
Description: To determine the effect of 2 weeks of treatment with inhaled montelukast plus mometasone and mometasone alone on bronchodilation assessed by average change from baseline in FEV1 over the 2 week treatment period; measurements taken at 1 and 2 weeks contributed to the average.
Time Frame: Baseline and 2 weeks
Population: The analysis was based on the Full analysis set (FAS) population which included all randomized patients who took at least one dose of blinded post randomization study drug (inhaled montelukast or matching placebo) and had a measurement for analysis available in at least one treatment period of the cross-over design.
Measure: Least Squares Mean (95% Confidence Interval); unit: L (Liter)
Groups:
- Montelukast + Mometasone: Inhaled montelukast 1mg (milligram) and open label mometasone 220 mcg (micrograms) once daily.
- Placebo + Mometasone: Inhaled placebo for montelukast and open label mometasone 220 mcg once daily.
Arm/Group | Montelukast + Mometasone | Placebo + Mometasone
Number analyzed (Participants) | 127 | 127
L (Liter) | 0.22 [0.15 to 0.30] | 0.17 [0.11 to 0.23]
Statistical Analysis 1: Comparison: Montelukast + Mometasone vs Placebo + Mometasone; Test type: Superiority or Other; p = 0.033, Mixed Models Analysis; Model with fixed effects for treatment, time (weeks 1 and 2), treatment-by-time interaction, period and baseline covariate; Difference in Least-Squares Means = 0.05, 95% CI [0.00 to 0.09] — Least-Squares Means for average change from baseline are derived using appropriate contrast from mixed model with fixed effects for treatment, time (weeks 1 and 2), treatment-by-time interaction, period and baseline covariate

2. Secondary Outcome: Change From Baseline in Daytime Asthma Symptom Score
Description: To determine the effect of 2 weeks of treatment with inhaled montelukast plus mometasone and mometasone alone on asthma symptoms assessed by average change from baseline in daytime asthma symptom score (which could range from 0 [best] to 6 [worst]) over the 2 week treatment period; measurements taken at 1 and 2 weeks contributed to the average.
Time Frame: Baseline and 2 weeks
Population: The analysis was based on the FAS population which included all randomized patients who took at least one dose of blinded post randomization study drug (inhaled montelukast or matching placebo) and had a measurement for analysis available in at least one treatment period of the cross-over design.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Montelukast + Mometasone | Placebo + Mometasone
Number analyzed (Participants) | 128 | 129
Units on a Scale | -0.39 [-0.49 to -0.29] | -0.24 [-0.35 to -0.12]
Statistical Analysis 1: Comparison: Montelukast + Mometasone vs Placebo + Mometasone; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least-Squares Means = -0.15, 95% CI [-0.26 to -0.05] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Nighttime Asthma Symptom Score
Description: To determine the effect of 2 weeks of treatment with inhaled montelukast plus mometasone and mometasone alone on asthma symptoms assessed by average change from baseline in nighttime asthma symptom score (which could range from 0 [best] to 3 [worst]) over the 2 week treatment period; measurements taken at 1 and 2 weeks contributed to the average.
Time Frame: Baseline and 2 weeks
Population: The analysis was based on a subset of the FAS population which included all randomized patients with nighttime symptoms at baseline (score>0), who took at least one dose of blinded post randomization study drug (inhaled montelukast or matching placebo) and had a measurement for analysis available in at least one treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Montelukast + Mometasone | Placebo + Mometasone
Number analyzed (Participants) | 89 | 90
Units on a Scale | -0.28 [-0.35 to -0.20] | -0.18 [-0.28 to -0.09]
Statistical Analysis 1: Comparison: Montelukast + Mometasone vs Placebo + Mometasone; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least-Squares Means = -0.09, 95% CI [-0.17 to -0.02] — [estimate comment as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Change From Baseline in Total Daily β-agonist Use
Description: To determine the effect of 2 weeks of treatment with inhaled montelukast plus mometasone and mometasone alone on as-needed β-agonist use assessed by average change from baseline in total daily β-agonist use over the 2 week treatment period; measurements taken at 1 and 2 weeks contributed to the average.
Time Frame: Baseline and 2 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs
Arm/Group | Montelukast + Mometasone | Placebo + Mometasone
Number analyzed (Participants) | 128 | 128
Puffs | -0.87 [-1.21 to -0.53] | -0.27 [-0.86 to 0.32]
Statistical Analysis 1: Comparison: Montelukast + Mometasone vs Placebo + Mometasone; Test type: Superiority or Other; p = 0.073, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least-Squares Means = -0.60, 95% CI [-1.26 to 0.06] — [estimate comment as in outcome 1, analysis 1]

5. Other Pre Specified Outcome: Percentage of Days With Asthma Control
Description: To determine the effect of 2 weeks of treatment with inhaled montelukast plus mometasone and mometasone alone on asthma control assessed by average percentage of days with asthma control over the 2 week treatment period; measurements taken at 1 and 2 weeks contributed to the average.
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Days
Arm/Group | Montelukast + Mometasone | Placebo + Mometasone
Number analyzed (Participants) | 129 | 129
Percentage of Days | 35.13 [28.52 to 41.74] | 29.04 [22.98 to 35.11]
Statistical Analysis 1: Comparison: Montelukast + Mometasone vs Placebo + Mometasone; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Model with fixed effects for treatment, time (weeks 1 and 2), treatment-by-time interaction and period; Difference in Least-Squares Means = 6.08, 95% CI [1.94 to 10.23] — Least-Squares Means for average percentage of days are derived using appropriate contrast from mixed model with fixed effects for treatment, time (weeks 1 and 2), treatment-by-time interaction and period

6. Other Pre Specified Outcome: Percentage of Days With Asthma Exacerbations
Description: To determine the effect of 2 weeks of treatment with inhaled montelukast plus mometasone and mometasone alone on worsening of asthma assessed by percentage of days with asthma exacerbations during the 2 week treatment period.
Time Frame: 2 Weeks
Population: The analysis was based on the Completers Set population which included all randomized patients who took a dose of blinded post randomization study drug (inhaled montelukast or matching placebo) in both treatment periods and had a measurement for analysis available in both treatment periods of the cross-over design.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Days
Arm/Group | Montelukast + Mometasone | Placebo + Mometasone
Number analyzed (Participants) | 127 | 127
Percentage of Days | 9.71 [5.51 to 13.90] | 15.14 [10.94 to 19.33]
Statistical Analysis 1: Comparison: Montelukast + Mometasone vs Placebo + Mometasone; Test type: Superiority or Other; p <= 0.001, ANCOVA; Model with terms for patient, treatment and period; Difference in Least-Squares Means = -5.43, 95% CI [-8.67 to -2.19] — Least-Squares Means for percentage of days are derived from ANCOVA model with terms for patient, treatment and period

7. Other Pre Specified Outcome: Change From Baseline in Total Peripheral Blood Eosinophils
Description: To determine the effect of 2 weeks of treatment with inhaled montelukast plus mometasone and mometasone alone on change from baseline in total peripheral blood eosinophils during the 2 week treatment period.
Time Frame: Baseline and 2 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^3/microliter
Arm/Group | Montelukast + Mometasone | Placebo + Mometasone
Number analyzed (Participants) | 119 | 119
10^3/microliter | -0.05 [-0.09 to -0.01] | 0.02 [-0.03 to 0.06]
Statistical Analysis 1: Comparison: Montelukast + Mometasone vs Placebo + Mometasone; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis; Model with fixed effects for treatment, period and baseline covariate; Difference in Least-Squares Means = -0.07, 95% CI [-0.12 to -0.01] — Least-Squares Means for change from baseline are derived from mixed model with terms for treatment, period and baseline covariate

8. Post Hoc Outcome: Change From Baseline in FEV1 (Forced Expiratory Volume; Volume of Air That is Exhaled During the First Second of a Forced Exhalation) in Patients Who Met Lung Function Eligibility Criteria Specifically at the Randomization Visit.
Description: To determine the effect of 2 weeks of treatment with inhaled montelukast plus mometasone and mometasone alone on bronchodilation assessed by average change from baseline in FEV1 over the 2 week treatment period in patients who met lung function eligibility criteria at randomization; measurements taken at 1 and 2 weeks contributed to average.
Time Frame: Baseline and 2 Weeks
Population: The analysis was based on a subset of the Full analysis set (FAS) population which included all randomized patients who took at least one dose of blinded post randomization study drug, had a measurement for analysis available in at least one treatment period and met lung function eligibility criteria specifically at the randomization visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: L (Liter)
Arm/Group | Montelukast + Mometasone | Placebo + Mometasone
Number analyzed (Participants) | 99 | 99
L (Liter) | 0.27 [0.19 to 0.35] | 0.19 [0.12 to 0.26]
Statistical Analysis 1: Comparison: Montelukast + Mometasone vs Placebo + Mometasone; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least-Squares Means = 0.08, 95% CI [0.03 to 0.13] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Groups:
- Montelukast + Mometasone: Inhaled montelukast 1 mg (milligram) and open label mometasone 220 mcg (micrograms) once daily.
Arm/Group | Montelukast + Mometasone | Placebo + Mometasone
Serious Adverse Events (participants affected / at risk) | 1/130 | 1/129
Other Adverse Events (participants affected / at risk) | 24/130 | 24/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast + Mometasone (N=130) | Placebo + Mometasone (N=129)
Pneumonia (Infections and infestations) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast + Mometasone (N=130) | Placebo + Mometasone (N=129)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Irritability (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 3
Pharyngitis (Infections and infestations) | 2 | 0
Pulpitis dental (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 1 | 2
Viral pharyngitis (Infections and infestations) | 0 | 1
Viral rhinitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 2 | 1
White blood cells urine positive (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 2
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.